CLINICAL TRIAL: NCT01773317
Title: Can Neuromuscular Training Alter Movement Patterns After Anterior Cruciate Ligament Injury?
Brief Title: Can Neuromuscular Training Alter Movement Patterns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lynn Snyder-Mackler (Other)
Responsible Party: Sponsor-Investigator, Lynn Snyder-Mackler, Principal Investigator, University of Delaware
Organization: University of Delaware (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 225014-1
Record Dates: First submitted 2012-06-13; First posted 2013-01-23 (Estimated); Last update posted 2019-07-25 (Actual); Status verified 2019-07

CONDITIONS: Acute Injury of Anterior Cruciate Ligament
MeSH Terms: interventions — Methods

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Perturbation (Experimental): Subjects complete the training protocol and peturbation training exercises
  Interventions: Other: Perturbation
- Control (Experimental): Subjects will complete the training protocol (including nordic hamstrings, standing squats, drop jumps, triple single leg hopping, and tuck jumps)
  Interventions: Other: Control

INTERVENTIONS:
Other: Perturbation — All subjects complete study protocol. Subjects randomized to the perturbation group will complete the additional perturbation exercises
  Other Names: Intervention
  Arms: Perturbation
Other: Control — Subjects will complete the study protocol (including nordic hamstrings, standing squats, drop jumps, triple single leg hopping, and tuck jumps)
  Other Names: Intervention
  Arms: Control

SUMMARY:
A prospective randomized controlled trial will be used to evaluate the efficacy of post-operative perturbation training. 80 patients who were regular participants in activities that involve cutting, pivoting, jumping, and lateral movements prior to injury who range in age from 13-55 at the time of injury are eligible. All eligible subjects must undergo primary anterior cruciate ligament reconstruction. Using a prospective randomized design, 40 subjects who will be block randomized by sex to 40 patients who will receive 10 sessions of post-operative perturbation training in addition to standard agility and return to activity progression and forty who receive only standard agility and return to activity progression. Post-operative perturbation training will be initiated when the athlete is at least 12 weeks post-anterior cruciate ligament reconstruction, has full range of motion and achieves 80% quadriceps strength symmetry, the criteria we currently use for beginning return to activity progression.

DETAILED DESCRIPTION:
For many years, our laboratory has been examining the functional capabilities and movement strategies of individuals who sustain anterior cruciate ligament injuries of the knee. Using a battery of clinical tests and measures with these athletes, we have learned that not all of these individuals respond similarly to injury. Some athletes, called potential copers, experience a high level of function after their injury. Rehabilitation that involves specialized training called perturbation training allows the majority of potential copers to be successful in returning to sports in the short-term. Non-copers, however, are a group of anterior cruciate ligament-injured athletes with poor knee stability during daily activities. The capability of these individuals to return to sport is limited, and anterior cruciate ligament reconstruction is typically recommended.

Over the last five years, we have begun to investigate the effects of perturbation training on non-copers. Non-copers represent the majority of anterior cruciate ligament-injured athletes, and they are of great interest not only because of their distinct functional limitations, but also the large variability within this group. Abnormal movement patterns are common following anterior cruciate ligament injury, but strategies differ between potential copers and non-copers. During an activity as basic as walking, non-copers reduce the motion of the injured knee and increase the work done at the hip and ankle, perhaps in an effort to avoid knee instability. Non-copers limit the motion of the knee by activating several muscles around the knee simultaneously. So while this may be effective in stabilizing the knee in the short term, this strategy may cause altered and potentially harmful loading patterns within the knee joint.

The abnormal movement and altered muscle firing patterns of anterior cruciate ligament-injured athletes are believed to be a mechanism for knee osteoarthritis. Though anterior cruciate ligament reconstruction restores knee stability, surgery does not fully address the faulty movement of these individuals. Pre-operative perturbation training is effective in improving function and normalizing knee motion in some non-copers. Perturbation training does not improve the ability of all non-copers to return to sport, suggesting other patient factors may be related to post-surgical outcomes. Women are known to be at greater risk for anterior cruciate ligament injury than men, but recently poorer outcomes in women following surgery have also been found. In response to pre-operative training, women demonstrate improved function and gait symmetry, but recover much more slowly after surgery and demonstrate abnormal patterns and knee joint loads. Persistent faulty patterns in women warrants further study and our research can help us find ways for us to address these abnormalities.

This goal of this work is to determine whether perturbation training can improve knee function and reduce faulty adaptations after anterior cruciate ligament reconstruction. Specifically, the aims of this project are to investigate whether the addition of post-operative perturbation training results in lower loading, better movement patterns and better functional outcomes than standard care.

ELIGIBILITY:
At this time, subjects have been enrolled and we are no longer recruiting for this study.

Inclusion Criteria:

* regular participants in activities that involve cutting, pivoting, jumping, and lateral movements prior to injury
* ages 13-55 at the time of injury
* undergo primary Anterior Cruciate Ligament reconstruction

Exclusion Criteria:

* concomitant Grade III ligament tears
* osteochondral defects >1cm2
* history of previous Anterior Cruciate Ligament Reconstruction or other major lower extremity injury/surgery

Ages: 13 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Actual)
Dates: Start 2011-11 (Actual); Primary Completion 2018-08-28 (Actual); Study Completion 2018-08-28 (Actual)

PRIMARY OUTCOMES:
Changes in gait patterns from baseline to completion of intervention (approximately 6 months after surgery), 1 year after anterior cruciate ligament reconstruction and 2 years after anterior cruciate ligament reconstruction | At enrollment (baseline), After protocol intervention (approximately 6 months after surgery), 1 year after anterior cruciate ligament reconstruction, 2 year after anterior cruciate ligament reconstruction
  Motion analysis data of gait patterns will be collected to analyze gait movement patterns of individuals after anterior cruciate ligament reconstruction and over time.

SECONDARY OUTCOMES:
Quadriceps Strength | At enrollment (baseline), After protocol intervention (approximately 6 months after surgery),1 year after anterior cruciate ligament reconstruction, 2 years after anterior cruciate ligament reconstruction
Patient reported outcomes (Knee Outcomes Survey-Activity of Daily Living Scale, Global Rating Score of Perceived Knee Function, Knee Injury and Osteoarthritis Outcome Score, International Knee Documentation Committee 2000 Subjective Knee Form) | At enrollment (baseline), After protocol intervention (approximately 6 months after surgery), 1 year after anterior cruciate ligament reconstruction, 2 years after anterior cruciate ligament reconstruction
Single-legged hop measures | At enrollment (baseline), After protocol intervention (approximately 6 months after surgery), 1 year after anterior cruciate ligament reconstruction, 2 years after anterior cruciate ligament reconstruction

CONTACTS AND LOCATIONS:
Overall Officials: Lynn Snyder-Mackler, PT,ATC,ScD, Principal Investigator — University of Delaware
Locations (1):
- University of Delaware, Physical Therapy Department, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ito N, Capin JJ, Khandha A, Buchanan TS, Silbernagel KG, Snyder-Mackler L. Bone-Patellar Tendon-Bone Autograft Harvest Prolongs Extensor Latency during Gait 2 yr after ACLR. Med Sci Sports Exerc. 2022 Dec 1;54(12):2109-2117. doi: 10.1249/MSS.0000000000003009. Epub 2022 Aug 6. PMID 35941514
- [Derived] Zarzycki R, Arhos E, Failla M, Capin J, Smith AH, Snyder-Mackler L. Association of the Psychological Response to the ACL-SPORTS Training Program and Self-reported Function at 2 Years After Anterior Cruciate Ligament Reconstruction. Am J Sports Med. 2021 Nov;49(13):3495-3501. doi: 10.1177/03635465211045388. Epub 2021 Oct 8. PMID 34623939
- [Derived] Capin JJ, Khandha A, Buchanan TS, Snyder-Mackler L. Partial medial meniscectomy leads to altered walking mechanics two years after anterior cruciate ligament reconstruction: Meniscal repair does not. Gait Posture. 2019 Oct;74:87-93. doi: 10.1016/j.gaitpost.2019.08.017. Epub 2019 Aug 27. PMID 31491565
- [Derived] Capin JJ, Failla M, Zarzycki R, Dix C, Johnson JL, Smith AH, Risberg MA, Huston LJ, Spindler KP, Snyder-Mackler L. Superior 2-Year Functional Outcomes Among Young Female Athletes After ACL Reconstruction in 10 Return-to-Sport Training Sessions: Comparison of ACL-SPORTS Randomized Controlled Trial With Delaware-Oslo and MOON Cohorts. Orthop J Sports Med. 2019 Aug 1;7(8):2325967119861311. doi: 10.1177/2325967119861311. eCollection 2019 Aug. PMID 31413963
- [Derived] Arundale AJH, Capin JJ, Zarzycki R, Smith A, Snyder-Mackler L. Functional and Patient-Reported Outcomes Improve Over the Course of Rehabilitation: A Secondary Analysis of the ACL-SPORTS Trial. Sports Health. 2018 Sep/Oct;10(5):441-452. doi: 10.1177/1941738118779023. Epub 2018 Jun 20. PMID 29924719
- [Derived] White K, Di Stasi SL, Smith AH, Snyder-Mackler L. Anterior cruciate ligament- specialized post-operative return-to-sports (ACL-SPORTS) training: a randomized control trial. BMC Musculoskelet Disord. 2013 Mar 23;14:108. doi: 10.1186/1471-2474-14-108. PMID 23522373